CLINICAL TRIAL: NCT00951236
Title: A Prospective, Randomized Study Comparing One vs. Two Cortisone Injections for Trigger Finger
Brief Title: Study Comparing One Versus Two Cortisone Injections for Trigger Finger
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Charles Leinberry, MD, Rothman Institute
Model: Parallel | Purpose: Treatment
Other Study IDs: RIUCLEI 09-01
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Stenosing Tenosynovitis; Trigger Finger
Keywords: Trigger Finger; Trigger Thumb
MeSH Terms: conditions — Tendon Entrapment; Trigger Finger Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One injection (Active Comparator)
  Interventions: Drug: One cortisone injection
- Two Injections (Active Comparator)
  Interventions: Drug: Two cortisone Injections

INTERVENTIONS:
Drug: One cortisone injection — Patients in this arm will receive one cortisone injection for the treatment of his/her symptoms
  Arms: One injection
Drug: Two cortisone Injections — Subjects randomized to this treatment will receive two cortisone injections, 4-6 weeks apart
  Arms: Two Injections

SUMMARY:
Trigger finger, also known as stenosing tenosynovitis, is a painful condition that can cause discomfort and disability. Many physicians choose to locally inject cortisone into the infected finger although there is no current consensus as to how many injections are needed to achieve maximum relief. This study will be a prospective, randomized study to compare one versus two injections for the treatment of trigger finger.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than 18 years of age, presenting with stenosing tenosynovitis.
* Subject is willing and able to provide informed consent.

Exclusion Criteria:

* Patients who have previously undergone surgery for the treatment of trigger finger.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2009-05

PRIMARY OUTCOMES:
To determine if there is a difference in the incidence of pain, stiffness, clicking or locking at 6 months following final injection

SECONDARY OUTCOMES:
To evaluate treatment response among diabetic patients
To evaluate treatment response between thumbs and fingers
To evaluate treatment response between nodular versus diffuse tenosynovitis

CONTACTS AND LOCATIONS:
Overall Officials: Charles Leinberry, MD, Principal Investigator — Rothman Institute; Pedro Beredjiklian, MD, Principal Investigator — Rothman Institute; Emran Sheikh, MD, Principal Investigator — Rothman Institute
Locations (7):
- United States (7):
  - Rothman Institute: Egg Harbor Township Location, Egg Harbor, New Jersey
  - Rothman Institute: Manahawkin location, Manahawkin, New Jersey
  - Rothman Institute: Vorhees location, Vorhees, New Jersey
  - Rothman Institute: Media location, Media, Pennsylvania
  - Rothman Institute Center City Location, Philadelphia, Pennsylvania
  - Rothman Institute, South Philadelphia Location, Philadelphia, Pennsylvania
  - Rothman Institute, Northeast Philadelphia location, Philadelphia, Pennsylvania